CLINICAL TRIAL: NCT01361386
Title: Long-Term Follow-up of Antithrombotic Management Patterns in Acute Coronary Syndrome Patients in Asia
Acronym: EPICOR ASIA
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CAP-XXX-2011/1
Record Dates: First submitted 2011-05-23; First posted 2011-05-26 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Acute Coronary Syndrome
Keywords: Long-term follow up; Antithrombotic management patterns; Acute Coronary Syndrome; Asia; quality of life
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
The purpose of this study is to describe the short-and long-tern (i.e. up to 2 years following the index event) AMPs in patients hospitalized for an acute coronary syndrome (i.e. STEMI or NSTE-ACS), and to document clinical outcomes, economic aspects and impact on quality of life of these AMPs in a 'real-life' setting.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent has been provided.
* Diagnosis of STEMI, NSTEMI or UA
* Hospitalization for the first time within 48 hours of onset of symptoms.

Exclusion Criteria:

* UA, STEMI, NSTEMI precipitated by or as a complication of surgery, trauma, or GI bleeding or post-PCI UA, STEMI and NSTEMI occurring in patients already hospitalized for other reasons.
* Current participation in a randomised interventional clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asian patients hospitalized for ACS within 48 hours of symptom onset and who have a final diagnosis of unstable angina (UA), STEMI or non-ST-segment elevation myocardial infarction (NSTEMI).
Sampling Method: Probability Sample
Enrollment: 13011 (Actual)
Dates: Start 2011-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
short- and long-term medication and treatment prescribed by physicians in real-life setting | up to 3 years

SECONDARY OUTCOMES:
clinical outcome (Cardiovascular events) | up to 3 years
cost of hospitalization | up to 3 years
quality of life (EQ-5D questionnaire) | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Guy Yeoman, Study Director — AstraZeneca; Prof. Huo Yong, Study Chair — Peking University 1st Hospital; Jayanti Visvanathan, Study Chair — AstraZeneca
Locations (108):
- China (45):
  - Research Site, Hefei, Anhui
  - Research Site, Wuhu, Anhui
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Chongqing, Chongqing Municipality
  - Research Site, Fuzhou, Fujian
  - Research Site, Lanzhou, Gansu
  - Research Site, Foshan, Guangdong
  - Research Site, Guangzhou, Guangdong
  - Research Site, Shenzhen, Guangdong
  - Research Site, Nanning, Guangxi
  - Research Site, Yulin, Guangxi
  - Research Site, Guiyang, Guizhou
  - Research Site, Baoding, Hebei
  - Research Site, Shijiazhuang, Hebei
  - Research Site, Tangshan, Hebei
  - Research Site, Daqing, Heilongjiang
  - Research Site, Harbin, Heilongjiang
  - Research Site, Zhengzhou, Henan
  - Research Site, Shiyan, Hubei
  - Research Site, Wuhan, Hubei
  - Research Site, Changsha, Hunan
  - Research Site, Nanjing, Jiangsu
  - Research Site, Wuxi, Jiangsu
  - Research Site, Xuzhou, Jiangsu
  - Research Site, Zhenjiang, Jiangsu
  - Research Site, Changchun, Jilin
  - Research Site, Jinzhou, Liaoning
  - Research Site, Shenyang, Liaoning
  - Research Site, Yingkou, Liaoning
  - Research Site, Xining, Qinghai
  - Research Site, Xi'an, Shaanxi
  - Research Site, Jinan, Shandong
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Changzhi, Shanxi
  - Research Site, Jinzhong, Shanxi
  - Research Site, Taiyuan, Shanxi
  - Research Site, Chengdu, Sichuan
  - Research Site, Tianjin, Tianjin Municipality
  - Research Site, Shihezi, Xinjiang
  - Research Site, Urumuqi, Xinjiang
  - Research Site, Kunming, Yunnan
  - Research Site, Hangzhou, Zhejiang
  - Research Site, Hong Kong
  - Research Site, Ningxia
  - Research Site, Qingdao
- India (26):
  - Research Site, Hyderabad, Andhra Pradesh
  - Research Site, Guwahati, Assam
  - Research Site, Ahmedabad, Gujarat
  - Research Site, Surat, Gujarat
  - Research Site, Vadodara, Gujarat
  - Research Site, Gurgaon, Haryana
  - Research Site, Bangalore, Karnataka
  - Research Site, Manipal, Karnataka
  - Research Site, Kochi, Kerala
  - Research Site, Trivandrum, Kerala
  - Research Site, Bhopal, Madhya Pradesh
  - Research Site, Bilāspur, Madhya Pradesh
  - Research Site, Aurangabad, Maharashtra
  - Research Site, Mumbai, Maharashtra
  - Research Site, Nagpur, Maharashtra
  - Research Site, Pune, Maharashtra
  - Research Site, Delhi, National Capital Territory of Delhi
  - Research Site, Ludhiana, Punjab
  - Research Site, Mohali, Punjab
  - Research Site, Ajmer, Rajasthan
  - Research Site, Jaipur, Rajasthan
  - Research Site, Chennai, Tamil Nadu
  - Research Site, Coimbatore, Tamil Nadu
  - Research Site, Madurai, Tamil Nadu
  - Research Site, Lucknow, Uttar Pradesh
  - Research Site, Kolkata, West Bengal
- Malaysia (2):
  - Research Site, Sarawak, Kuching
  - Research Site, George Town
- Research Site, Singapore, Singapore
- South Korea (12):
  - Research Site, Busan, Busan
  - Research Site, Chuncheon, Chuncheon
  - Research Site, Cheonan, Chungcheongnam-do
  - Research Site, Deagu, Deagu
  - Research Site, Gwangju, Gwangju
  - Research Site, Bucheon-si, Gyeonggi-do
  - Research Site, Goyang-si, Gyeonggi-do
  - Research Site, Suwon, Gyeonggi-do
  - Research Site, Yangsan, Gyeongsangnam-do
  - Research Site, Jeju City, Jeju-do
  - Research Site, Iksan, Jeollabuk-do
  - Research Site, Seoul, Seoul
- Thailand (20):
  - Research Site, Bangkoknoi, Bangkok
  - Research Site, Huaykwang, Bangkok
  - Research Site, PathumWan, Bangkok
  - Research Site, Payathai, Bangkok
  - Research Site, Rachathevi, Bangkok
  - Research Site, Saimai, Bangkok
  - Research Site, Muang, Changwat Chanthaburi
  - Research Site, Muang, Changwat Chon Buri
  - Research Site, Muang, Changwat Lampang
  - Research Site, Muang, Changwat Nan
  - Research Site, Klongluang, Changwat Pathum Thani
  - Research Site, Muang, Changwat Phitsanulok
  - Research Site, Muang, Changwat Songkhla
  - Research Site, Muang, Changwat Suphan Buri
  - Research Site, Muang, Changwat Surat Thani
  - Research Site, Muang, Chiangmai
  - Research Site, Muang, Chiangrai
  - Research Site, Muang, Khonkaen
  - Research Site, Muang, Nakornratchaseema
  - Research Site, Muang, Udonthani
- Vietnam (2):
  - Research Site, Ho Chi Minh City, Ho Chi Minh City
  - Research Site, Huế, Hue

REFERENCES:
- [Derived] Huo Y, Van de Werf F, Han Y, Rossello X, Pocock SJ, Chin CT, Lee SW, Li Y, Jiang J, Vega AM, Medina J, Bueno H. Long-Term Antithrombotic Therapy and Clinical Outcomes in Patients with Acute Coronary Syndrome and Renal Impairment: Insights from EPICOR and EPICOR Asia. Am J Cardiovasc Drugs. 2021 Jul;21(4):471-482. doi: 10.1007/s40256-020-00447-5. Epub 2021 Feb 4. PMID 33537947
- [Derived] Guan S, Xu X, Li Y, Li J, Guan M, Wang X, Jing Q, Huo Y, Han Y. Impact of Diabetes Mellitus on Antithrombotic Management Patterns and Long-Term Clinical Outcomes in Patients With Acute Coronary Syndrome: Insights From the EPICOR Asia Study. J Am Heart Assoc. 2020 Nov 17;9(22):e013476. doi: 10.1161/JAHA.119.013476. Epub 2020 Nov 7. PMID 33164633
- [Derived] Zhang S, Wang W, Sawhney JPS, Krittayaphong R, Kim HS, Nhan VT, Lee SW, Ong TK, Chin CT, Pocock SJ, Huo Y, Qian J, Ge J. Antithrombotic management and long-term outcomes following percutaneous coronary intervention for acute coronary syndrome in Asia. Int J Cardiol. 2020 Jul 1;310:16-22. doi: 10.1016/j.ijcard.2020.01.008. Epub 2020 Mar 17. PMID 32192746
- [Derived] Jan S, Lee SW, Sawhney JPS, Ong TK, Chin CT, Kim HS, Krittayaphong R, Nhan VT, Pocock SJ, Vega AM, Hayashi N, Huo Y. Predictors of high-cost hospitalization in the treatment of acute coronary syndrome in Asia: findings from EPICOR Asia. BMC Cardiovasc Disord. 2018 Jul 4;18(1):139. doi: 10.1186/s12872-018-0859-4. PMID 29973147